CLINICAL TRIAL: NCT02821390
Title: Analgesic Effect Of Topical Nepafenac 0.1% On Pain Related To Intravitreal Injections: A Randomized Crossover Study
Brief Title: Effect of Topical Nepafenac 0.1% on Pain Related to Intravitreal Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Constantinos D. Georgakopoulos, MD, PhD, Assoc. Professor, University Hospital of Patras
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 72/15.04.16
Record Dates: First submitted 2016-06-27; First posted 2016-07-01 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Pain
Keywords: intravitreal injection; pain; non-steroidal anti-inflammatory drugs; anti-VEGF; nepafenac
MeSH Terms: conditions — Pain | interventions — nepafenac; Ophthalmic Solutions; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nepafenac 0.1% Eye Drops (Active Comparator): One drop of Nepafenac 0.1% Eye Drops will be instilled to the eye's cul de sac prior to the intravitreal injection.
  Interventions: Drug: Nepafenac Eye Drops
- Artificial Tears (Placebo Comparator): One drop of Artificial Tears will be instilled to the eye's cul de sac prior to the intravitreal injection.
  Interventions: Drug: Placebo (Artificial Tears)

INTERVENTIONS:
Drug: Nepafenac Eye Drops — One drop instilled to the eye's cul de sac prior to the intravitreal injection.
  Other Names: NEVANAC 0.1% Eye Drops
  Arms: Nepafenac 0.1% Eye Drops
Drug: Placebo (Artificial Tears) — One drop instilled to the eye's cul de sac prior to the intravitreal injection
  Other Names: TEARS NATURALE 0.1%+0.3% Eye Drops
  Arms: Artificial Tears

SUMMARY:
The analgesic effect of Nepafenac 0.1% Ophthalmic Drops on ocular pain related to intravitreal injections will be evaluated.

Pain perception will be assessed by the Short Form of the McGill Pain Questionnaire.

DETAILED DESCRIPTION:
Intravitreal injection (IVI) is a preferred route of administration of drugs in the posterior segment of the eye. Intravitreal injection of anti-VEGFs constitutes the mainstay for the treatment of various retinal diseases such as AMD, RVO, DME etc.

The procedure of the IVI is, however, associated with a level of discomfort for the patient.

Ophthalmic nonsteroidal anti-inflammatory drugs (NSAIDs) constitute an established and effective treatment option for the management of inflammation and pain associated with cataract surgery and of pain associated with corneal refractive surgery, for inhibition of intraoperative miosis and for the treatment of seasonal allergic conjunctivitis.

The primary goal of this study is to assess the analgesic effect of Nepafenac 0.1% Eye Drops a topical NSAID on pain related to intravitreal injections immediately after and up to six hours post-IVI.

A number of patients scheduled to undergo IVIs will be divided in two groups. All patients must have already undergone at least one IVI. In patients receiving IVIs in both eyes only one eye will be included in the study.

The patients of the first group will be randomized to receive Nepafenac 0.1% Eye Drops in the first appointment and then crossover to receive the placebo (Artificial Tears) in their next appointment for an IVI.

The patients of the second will be randomized to receive the placebo (Artificial Tears) in the first appointment and then crossover to receive Nepafenac 0.1% Eye Drops in their next appointment for an IVI.

All drugs will be administered prior to the injection by a member of the Department's personnel (a staff nurse).

Patients will be required to complete the greek version of the short form McGill Pain Questionnaire (SF-MPQ) comprising of the Visual Analogue Scale, the main component of the SF-MPQ and the Present Pain Intensity Scale immediately after the injection and 6 hours post-IVI.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be patients of the Medical Retina Department of our Clinic, who are scheduled to receive IVIs of ranibizumab (Lucentis; Novartis Pharma S.A.S., Huningue, France) or aflibercept (Eylea; Bayer Healthcare Pharmaceuticals, Berlin, Germany) in one eye and had already undergone at least one IVI of an anti-VEGF agent.

Exclusion Criteria:

* History of previous eye surgery other than cataract extraction surgery, herpetic eye disease, uncontrolled glaucoma, uveitis, active conjunctivitis, keratitis and bullous keratopathy, a previously known allergic response to bromfenac or other NSAIDs and salicylates, any systemic or topical use of NSAIDs or any use of sedative medications within 7 days from the visit and during the day of IVI.
* Patients with poor cooperation in understanding and answering the questions of the SF-MPQ, including the visual analogue scale (VAS).
* Unsuccessful blinding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Nepafenac's analgesic effect in patients undergoing intravitreal injections of anti-VEGFs as measured by the Visual Analogue Scale. | Immediately and 6 hours after injection

SECONDARY OUTCOMES:
Assessment of Nepafenac's analgesic effect after intravitreal injections of anti-VEGFs as measured by the main component of the short form of the McGill Pain Questionnaire | Immediately and 6 hours after injection
Assessment of Nepafenac's analgesic effect after intravitreal injections of anti-VEGFs as measured by the main component of the Present Pain Intensity score | Immediately and 6 hours after injection

CONTACTS AND LOCATIONS:
Overall Officials: Constantine D Georgakopoulos, MD, Phd, Principal Investigator — Associate Professor of Ophthalmology, Medical School, University of Patras, Greece
Locations (1):
- University Hospital of Patras, Pátrai, Achaea, Greece

IPD SHARING:
Plan to Share IPD: Undecided